CLINICAL TRIAL: NCT01723995
Title: Effect of Low-level of Laser Therapy in Nipple Trauma During Breastfeeding
Brief Title: Laser Therapy in Nipples Injured During Breastfeeding
Acronym: LTNIBF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Kelly Pereira Coca, PhD student - Nurse midwife, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEP 1710-9
Record Dates: First submitted 2012-10-10; First posted 2012-11-08 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Nipple Trauma
Keywords: nipple/injure; breastfeeding; pain; laser
MeSH Terms: conditions — Breast Feeding; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- low-level laser on nipples (Experimental): Application of laser light from the device in direct contact with the nipple injury, equipment connected and set up at a dose of 5J/cm2 (Epoint = 0.2J/cm2) for both groups, three consecutive doses of 5J/cm2 (ETotal = 0.6J/cm2) along the entire length of the injury.
  Interventions: Radiation: low-level laser on nipples
- low-level laser off on nipples (Placebo Comparator): Laser with modified standard operation - shutdown of InGaAIP semiconductor diode and installation of a visible red light emitting diode with optical power of 0mW (LED - Light Emitting Diode - maximum power with standard nozzle).
  Interventions: Radiation: low-level laser on nipples

INTERVENTIONS:
Radiation: low-level laser on nipples — The LASER HAND WL device, manufactured by MM Optics.
  Other Names: LASER HAND WL InGaAIP semicondutor; registered by ANVISA/MS No. 80051420009; wavelength 660 nn; Optical power 40mW; visible red spectrum range; with emission of continuous light (CW)

SUMMARY:
This study aims to evaluate the effect of low-level laser in pain relief and tissue repair in mothers with nipple trauma during breastfeeding, compared to a control group.

DETAILED DESCRIPTION:
The selection was made through the search of women hospitalized in Accommodation beds with nipple trauma, lifting of stipulated criteria, and inclusion of women in the study upon acceptance and signing of the consent form. To collect the data, a group was formed with people trained as evaluators, responsible for election, randomization, filling of First Assessment and Subsequent Assessment forms, recording of photo images and pain evaluation before and after treatment with laser; and applicators, responsible for laser handling and irradiation. Data collection followed the following order: filling of the first instrument, breast image capture, suckling observation, identification of pain during the child's breast sucking, laser irradiation and re-identification of pain during the child's breast sucking after laser treatment. The collection of data of this form occurred continuously every twelve hours until repair of the nipple trauma or patient discharge. A minimum of two and a maximum of six assessments were carried out, from the inclusion of the patient in the study (taken as zero hour) to 60 hours postpartum. Irradiation, in turn, was performed every 24 hours during the same period, including one to three irradiations per patient in each of the breasts.

ELIGIBILITY:
Inclusion Criteria:

Women hospitalized in the Accommodation System with their children, feeding exclusively directly from the breast and presenting unilateral or bilateral nipple trauma.

Exclusion Criteria:

Women who were using any other form of treatment for nipple trauma; use of any topical substance in the nipple-areola region; presence of inverted and pseudo-inverted nipple; presence of mastitis; previous history or presence of malignancies; presence of photosensitivity or any adverse reactions to exposure to sunlight; discharge planned for the first day of data collection; women under unfavorable psycho-affective and cognitive situations which prevented assessment of the analog pain scale, photo image record. and observation of breastfeeding; women who had twins, children with gestational age less than 37 weeks, or birth weight less than 2500 grams.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2011-02; Primary Completion 2011-11 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Reduction of nipple pain during breastfeeding | Time - between 12 and 60 hours
  The mothers treated with low-level laser therapy should present a decrease in the degree of pain during breastfeeding in the presence of nipple trauma compared to the control group.

SECONDARY OUTCOMES:
Tissue repair in nipples during breastfeeding | Between 12 and 60 hours
  Secondarily, the nipple wound characteristics shall be assessed regarding tissue repair with the use of laser, compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly P. Coca, MD, Principal Investigator — Student - Federal University of Sao Paulo; Ana CV Abrão, PHD, Principal Investigator — Federal University of São Paulo; Monica A. Gamba, PHD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo - Sao Paulo School of Nursing, São Paulo, Brazil